CLINICAL TRIAL: NCT06137924
Title: Intraoperative Autonomic Neural Blockade (ANB) Comparison Between Different Local Anesthetic Combinations. A Randomized Clinical Trial Protocol
Brief Title: Intraoperative Autonomic Neural Blockade
Acronym: ANB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Simón Bolívar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PRO-CEI-USB-CE-0394-02
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative; Nausea, Postoperative; Vomiting, Postoperative; Analgesia; Opioid Use
Keywords: autonomic neural blockade; visceral pain; postoperative nausea and vomiting; opioids
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Agnosia; Visceral Pain | interventions — Dexamethasone; Clonidine

STUDY DESIGN:
Intervention Model Description: Three arms using different local anesthetic combinations: bupivacaine plus dexamethasone, bupivacaine plus dexamethasone and a plasma substitute and bupivacaine plus clonidine.
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed using sealed envelopes stratified by the institution in blocks of six. The data manager will prepare these envelopes. The data manager will store the randomization list containing the final treatment assignments. Only the data manager will have access to the randomization list throughout the study. These sealed envelopes will be placed in the patient's chart and will not be opened until the patient is in the operating room and general anesthesia has been initiated. The patient and the independent investigator assessing and recording the patient's data will be masked to treatment arm assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ANB with 0.5% bupivacaine plus dexamethasone 8 mg (Active Comparator): ANB will be performed using 5% bupivacaine 20 cc plus dexamethasone 8 mg as the local anesthetic.
  Interventions: Drug: Local anesthetic injection Bupivacaine plus dexamethasone
- ANB with 0.5% bupivacaine plus dexamethasone and a colloid (Experimental): ANB will be performed in this group using 0.5% bupivacaine 20 ccs plus dexamethasone 8 mg and a plasma volume substitute (succinylated gel).
  Interventions: Drug: Local anesthetic injection bupivacainde plus dexamethasone plus a colloid
- 0.5% bupivacaine plus clonidine 0.145 mcg (Experimental): ANB with will be performed in this group using 0.5% bupivacaine 20 ccs plus clonidine 0.145 mcg.
  Interventions: Drug: Local anesthetic injection bupivacaine plus clonidine

INTERVENTIONS:
Drug: Local anesthetic injection Bupivacaine plus dexamethasone — The autonomic neural block is performed with a 25-gauge needle attached to a venous catheter extension introduced through the left 12-mm port. Infiltration of 20 mL of non-diluted 0.5% bupivacaine plus dexamethasone 8 mg is performed at the celiac plexus and vagus nerve trajectory.
  Arms: ANB with 0.5% bupivacaine plus dexamethasone 8 mg
Drug: Local anesthetic injection bupivacainde plus dexamethasone plus a colloid — bupivacaine plus dexamethasone 8 mg plus a colloid 10 cc (Gelofucin, B. Braun Medical S.A., Crissier, Suiza.) is performed at the celiac plexus and vagus nerve trajectory.
  Arms: ANB with 0.5% bupivacaine plus dexamethasone and a colloid
Drug: Local anesthetic injection bupivacaine plus clonidine — bupivacaine 5% plus clonidine (0,150mgs) is performed at the celiac plexus and vagus nerve trajectory
  Arms: 0.5% bupivacaine plus clonidine 0.145 mcg

SUMMARY:
The duration of the effect of autonomic neural blockade (ANB) is the most critical limitation for successful clinical application. The analgesic effect using only 0.5% bupivacaine may wear off after 12 to 18 hours. We have prolonged this effect using a combination of bupivacaine and dexamethasone. In this protocol, we aim to study three different local anesthetic combinations to prolong the effect of the ANB.

DETAILED DESCRIPTION:
The study described herein is a prospective, double-blinded RCT involving patients undergoing laparoscopic sleeve gastrectomy (LSG) at Clínica Portoazul and Clínica Iberoamérica in Barranquilla, Colombia. The patients will be randomized to one of three parallel groups: ANB using 5% bupivacaine plus dexamethasone, 5% bupivacaine plus dexamethasone and a colloid, and 5% bupivacaine plus clonidine.

Patients All adult patients scheduled for LSG at each participating institution will be eligible for screening for study inclusion and granting of consent to study participation. The exclusion criteria will be the inability to perform an ANB because of anatomical difficulties, the need for revisional surgery, the need for concurrent surgical procedures beyond hiatal hernia repair, conversion to open surgical procedures, allergies to local anesthetics, and intraoperative complications (e.g., visceral or vascular perforations, or anesthesia-related complications requiring admission to intensive care).

Sample size The estimated sample size in each group was 50 patients ( total enrollment of 150 patients), assuming that for a balanced one-way ANOVA, using a sample size of 120 (each group: 40) would provide a statistical power of 0.9, with a significant level of 0.01 and a standard deviation of 3.

ANB The autonomic neural block is performed with a 25-gauge needle attached to a venous catheter extension introduced through the left 12-mm port. The needle is capped during its introduction, and the cap is removed inside the abdomen using a grasper and kept under direct vision. Infiltration of 20 mL of non-diluted 0.5% bupivacaine plus dexamethasone 8 mg, bupivacaine plus dexamethasone 8 mg plus a colloid 10 cc (Gelofusin, B. Braun Medical S.A) or bupivacaine 5% plus clonidine (0,150mgs) is performed at six levels with careful aspiration preceding fluid infiltration. After elevating the stomach with a grasper at the most proximal aspect of the lesser curvature and creating two windows at each side of the verticalized left gastric artery, two of the infiltrations are performed at t the base of the left gastric artery (Fig. 2). Four areas are infiltrated at the track of vagus nerves and branches. ANB is reinforced at the final stage of the procedure. When initial exposure of the celiac trunk proved difficult, elevating the sleeve can facilitate the procedure. The procedure is rapid, reproducible, and proven safe in a previous RCT. However, it has a learning curve. Details of the procedure are available.

Data collection An independent investigator will be responsible for collecting and recording the study data. Patients' age, sex, body mass index, current medications, and medical and surgical history will be recorded prospectively with informed consent at their visit to the preoperative clinic at the time of study enrollment. Details of the procedure will be consigned in the surgical record. An analog pain scale survey is administered by an investigator blinded to the patients' groups in person at one hour (in the recovery room), eight hours postoperatively the following morning, and by phone at 36 hours. The investigator recorded the need for analgesics and the presence of nausea, vomiting, and other symptoms at the same periods.

Statistical analysis Continuous outcome variables will be compared with two-sample t-tests. Categorical and binary outcome variables will be compared using chi-squared tests.

Analgesia protocol All patients received proton pump inhibitors, conventional antiemetics, and a scheduled baseline analgesic such as acetaminophen (1 g intravenously every six h) or dipyrone (1 g intravenously every six h). A nonsteroidal anti-inflammatory drug such as diclofenac and hyoscine butyl bromide (0.2 mg intravenously) is administered in non-allergic patients 12 14 hours post-surgery and the following morning if necessary. The rescue analgesic was Oxycodone (3 mg every 6 h). Oxycodone was the only opioid derivative used. After surgery, a popsicle was offered in the afternoon, and clear fluids were started the following day. Patients are discharged from the hospital in the afternoon the next day after surgery if they are hemodynamically within normal limits, tolerate clear fluids, and have controlled pain.

ELIGIBILITY:
Inclusion Criteria:

All adult patients scheduled for Laparoscopic Sleeve Gastrectomy(LSG) at each participating institution will be eligible for screening for study inclusion and granting of consent to study participation.

Exclusion Criteria:

The exclusion criteria will be the inability to perform an ANB because of anatomical difficulties, the need for revisional surgery, the need for concomitant surgical procedures beyond hiatal hernia repair, conversion to open surgical procedures, allergies to local anesthetics, and intraoperative complications (e.g., visceral or vascular perforations, or anesthesia-related complications requiring admission to intensive care).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-02 (Estimated); Primary Completion 2024-04-02 (Estimated); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | measured at 1,8,24 and 36 hours after surgery
  pain will be measured using an analog visual scale 0-10 being o no pain and 10 the most excruciating pain.

SECONDARY OUTCOMES:
nausea | at 1,8,24 and 36 hours after surgery
  the presence of postoperative nausea will be determined.
vomiting | at 1,8,24 and 36 hours after surgery.
  The presence of postoperative vomiting will be determined.
total doses of analgesics beyond the basic analgesic protocol. | at 1,8,24 and 36 hours after surgery.
  total doses of any analgesic needed beyond the basic protocol
total doses of opioids required | at 1,8,24 and 36 hours after surgery
  total doses of opioids required
level of pain in the subgroup of patients with hiatal hernia repair | at 1, 8, 24 and 36 hours after surgery
  To establish the level of pain using the analog visual scale in the subgroup of patients that requiered a hiatal hernia repair beyond the basic procedure (laparsocopic sleeve gastrectomy)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daes J, Morrell DJ, Hanssen A, Caballero M, Luque E, Pantoja R, Luquetta J, Pauli EM. Paragastric Autonomic Neural Blockade to Prevent Early Visceral Pain and Associated Symptoms After Laparoscopic Sleeve Gastrectomy: a Randomized Clinical Trial. Obes Surg. 2022 Nov;32(11):3551-3560. doi: 10.1007/s11695-022-06257-9. Epub 2022 Sep 2. PMID 36050617
- [Background] Daes J, Pantoja R, Luquetta J, Luque E, Hanssen A, Rocha J, Morrell DJ. Impact on Anesthetic Agent Consumption After Autonomic Neural Blockade as Part of a Combined Anesthesia Protocol: A Randomized Clinical Trial. Anesth Analg. 2024 Sep 1;139(3):581-589. doi: 10.1213/ANE.0000000000006769. Epub 2023 Dec 13. PMID 38091501
- [Background] Daes J, Rocha J, Luque E, Hanssen A. Comparative effectiveness of bupivacaine- dexamethasone and liposomal bupivacaine for autonomic neural blockade in laparoscopic sleeve gastrectomy: a study on pain, postoperative nausea and vomiting and analgesic consumption. British journal of surgery. Abstract presented at 2023 IBC-University of Oxford World Congress; British Journal of Surgery Oral Abstract Prize Session. Oxford University; London, UK. September 20, 2023. Forthcoming 2023.
- [Derived] Daes J, Pantoja R, Luque E, Hanssen A, Rocha J, Pauli EM. Intraoperative autonomic neural blockade: comparison between different local anesthetics combinations: a randomized clinical trial. Surg Endosc. 2025 Apr;39(4):2523-2533. doi: 10.1007/s00464-025-11637-0. Epub 2025 Mar 3. PMID 40032662